CLINICAL TRIAL: NCT06659497
Title: The Level of Infertility Distress and Fertility Readiness of Women Receiving Web-Based Education on the Treatment Process: A Randomised Controlled Study
Brief Title: The Level of Infertility Distress and Fertility Readiness of Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, Hilal Karadeniz, Research Assistant Phd, Duzce University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/50
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Infertility; Intrauterine Insemination (IUI)
Keywords: Intrauterine insemination; infertility; nursing education; web based education
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: The research is being conducted as a randomized controlled experimental study to determine the effects of web-based training on the treatment process of women undergoing Intrauterine Insemination (IUI) treatment on the level of infertility, fertility readiness and pregnancy outcomes. There are 2 groups of subjects in the study as experimental and control. Block randomization was applied in determining the groups. In this direction, the following randomization steps were followed by the statistics expert in order to eliminate bias and increase the reliability of the study. Randomization was done according to the educational status of the women (primary school - secondary school, high school, university and above when grouped) in a way that homogeneity was ensured in each group and it was planned to be statistically re-evaluated at the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Patients in this group participate in a web-based training application. Patients are asked pre-test questions before the training and pre-test questions after the training.
  Interventions: Behavioral: web-based patient education
- Control (No Intervention): No intervention is made for patients in this group. Patients are asked pre-test questions before treatment and pre-test questions after treatment.

INTERVENTIONS:
Behavioral: web-based patient education — The web-based training, which will provide the following information about the IUI treatment process, will last a total of 60 minutes.
  MODULE 1: General Information About Fertility MODULE 2: Diagnostic and Therapeutic Methods in Infertility / Insemination Treatment MODULE 3: Drugs Used in Insemination Treatment and Their Application MODULE 4: Things to Consider After Insemination
  Arms: intervention

SUMMARY:
The infertility treatment process is a multidisciplinary teamwork involving different professional groups. Especially the Controlled Ovarian Hyperstimulation (COH) protocols applied during the infertility treatment process require good nursing education, close monitoring and effective counseling. The patient's education during this process, the development of self-administration skills and follow-up are the responsibility of the infertility nurse and directly affect the treatment process and its success. There is a need to determine the level of impact of infertile individuals on this process, to increase their knowledge level regarding the treatment process and to ensure that individuals are supported closely and strengthened during the treatment process. This study was planned as a randomized controlled experimental study to determine the effect of web-based training to be given to women who undergo Intrauterine Insemination (IUI) treatment on the level of impact of infertility and fertility readiness of women.

DETAILED DESCRIPTION:
Infertility is defined as the failure of couples of reproductive age to conceive or to continue a pregnancy despite having unprotected sexual intercourse at least twice a week for a year. When we look at infertility rates worldwide, it is thought that more than 80 million people cannot have children due to medical reasons, and in Turkey, an average of 15% of couples are diagnosed with infertility. Although infertility is not a life-threatening problem, it is often considered a stressful life event for couples or individuals due to the meaning that individuals or society attribute to having children. At the same time, it is a condition that brings medical, physiological, psychological and social problems, has cultural, religious and class aspects, confronts the individual with unexpected stressors, and changes the couple's quality of life. For all these reasons, the diagnosis of infertility creates a crisis in couples that they do not know how to cope with. Many studies revealing the psychological dimensions of infertility and assisted reproductive treatments have shown that infertility negatively affects individuals by causing an increase in their stress, depression and anxiety levels. Readiness is the person's evaluation of their own abilities and situation, considering existing options, producing and implementing new solutions. A high level of readiness encourages individuals to experience psychological reactions such as anger and depression less and to have a more positive approach. A lower level of readiness can cause individuals to feel depressed, afraid and vulnerable in the face of change. The level of fertility readiness, which is affected by social, economic and personal factors, is similarly linked to perceived abilities for parenting. This situation also affects fertility treatment, and it is reported that as the level of feeling ready for fertility treatment increases, treatment results are also positive. Web-based education is an internet-based distance education model that increases the quality of education services today. Studies indicate that web-based education is important in terms of eliminating physical or spatial distances and thus enabling individuals in geographically different places to easily access educational resources. In addition, web-based education offers the opportunity to access educational materials at the time and frequency desired by the participant. It allows the participant to control the pace of the training and to reinforce their knowledge with the opportunity to repeat the training when necessary, and to make the training effective and permanent. The infertility treatment process is a multidisciplinary team effort involving different professional groups. Especially the Controlled Ovarian Hyperstimulation (COH) protocols applied during the infertility treatment process require good nursing education, close monitoring and effective consultancy. The infertility nurse is responsible for educating the patient during this process, developing their self-application skills and monitoring them, and this directly affects the treatment process and its success. There is a need to determine the level of infertile individuals being affected by this process, to increase their knowledge level regarding the treatment process, and to ensure that individuals are closely supported and strengthened during the treatment process. This study was planned as a randomized controlled experimental study in order to determine the effect of web-based education to be given to women undergoing Intrauterine Insemination (IUI) treatment on the level of infertility and fertility readiness of women. In this way, it is thought that in addition to face-to-face nursing education and counseling given to female patients in infertility treatment, the usability of web-based education in this field can be evaluated, the effectiveness and quality of education can be increased by integrating web-based education into the process, the close and continuous follow-up of patients can be ensured, possible incorrect treatment process management can be prevented, and the couple can be prevented from being negatively affected by this process both materially and morally by preventing cycle losses.

The study was planned to be conducted between 15.03.2024 and 15.12.2024 on women between the ages of 18-45 who applied to Düzce University Health Application and Research Center, Infertility Polyclinic.The study universe consists of all women who applied to Düzce University Health Application and Research Center, Infertility Polyclinic between 15.03.2024 and 15.08.2024 and met the inclusion criteria. Study sample; Based on a similar study conducted previously, the Power analysis (G*Power 3.1.9.2) was performed, and the effect size was determined as 0.61, the power as 80%, and the α-type error estimate as 0.05, and the sample size for each group was determined as 34 infertile women. The drop-out number (the number of those who did not continue the study) was taken as 5, and the sample size was determined as 39 for each group. In the study, 45 patients will be tried to be reached in each group, including the experimental and control groups, considering possible data losses. Block randomization will be applied in determining the groups.Data will be collected using the Personal Information Form, Infertility Impact Scale (IAS) and Fertility Readiness Scale for Women Receiving Fertility Support.

A preliminary application will be conducted to evaluate the understandability and usability of the Personal Information Form developed by the researchers by the individuals in the sample group. For this purpose, an average of 9 women, who constitute 10% of the 90-person sample determined according to the calculation of the minimum sample number to be reached in the place where the research will be conducted, will be included in the preliminary application. After the preliminary application, the data collection form will be finalized and the data collected for the preliminary application will not be included in the research.

Research data will be collected between 15.03.2022-15.12.2023. The collection of research data will be completed within approximately 20 days for each patient from the beginning of the KOH treatment to pregnancy determination for patients scheduled for Controlled Ovarian Hiperstimulation (KOH) during the Intrauterine Insemination (IUI) treatment process. Before starting the research, women in the experimental and control groups who applied to the infertility clinic and met the inclusion criteria for the research will be interviewed face to face and informed about the purpose, duration, planned flow and the contribution that the research application can make to the treatment process will be provided, and verbal consent will be obtained from women who agree to participate in the research. Then, contact information (name, surname, telephone number, Turkish ID number) of all patients in the randomized experimental and control groups will be collected and user registrations will be completed in order to provide access to the website via www.asilamatedavisi.com only for women in the experimental group. The women in both groups will fill out the Personal Information Form, pre-test forms and the post-test forms within 1 week after the vaccination process, by reaching them through the survey link (Google forms) that will be prepared online. During the data collection phase, participants will be able to participate in the study after reading and approving the informed consent form that appears before they can access the questionnaires prepared via Google Forms. Filling out the questionnaires will take approximately 15-20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Those who applied to Düzce University Health Application and Research Center Infertility Polyclinic between 15.03.2024-15.08.2024,
* Primary infertility,
* Those who are planned to use Controlled Ovarian Hyperstimulation (COH) in intrauterine insemination (IUI) treatment,
* Those who have the equipment (mobile phone, computer, tablet, internet, etc.) to access web-based education,
* Those who do not have a chronic disease,
* Those who do not have a diagnosed psychiatric disease,
* Those who agree to participate in the study,
* Those who have the ability to understand and comprehend the questionnaires

Exclusion Criteria:

* Those who are not planned to use Controlled Ovarian Hyperstimulation (COH) in intrauterine insemination (IUI),
* Those who give up on treatment,
* Those who have 3 or more graff follicle development on the day of insemination (treatment cancellation),
* Those who have 1 million or less sperm obtained on the day of insemination (treatment cancellation)

Ages: 23 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The research is conducted only with infertile women
Enrollment: 90 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Level of Infertility Affectedness | up to 5 months
  In the research, the level of women's impact on infertility is measured with a Infertility Distress Scale.
  Infertility Distress Scale: The scale defines how people's cells and emotional states continue to be affected by infertility. The scale consists of a total of 21 items, 16 of which are direct and five are reverse. Reverse items are items 3, 10, 13, 14 and 21. The scale is a 4-point Likert type and positive items are scored as 1: never, 4: always, while negative items are scored the opposite way. A score between 21 and 84 is obtained from the scale. There is no cut-off score for the scale. High scores obtained from the scale indicate that the effect of infertility is high. In addition, there is no subscale of the operation. The reliability of the item scores of the scale is applied as 0.93.

SECONDARY OUTCOMES:
Fertility Readiness | up to 5 months
  In the research, women's level of readiness for pregnancy is measured with a Fertility Readiness Scale for Women Receiving Fertility Support scale.
  Fertility Readiness Scale for Women Receiving Fertility Support: The scale is used for women who want to become pregnant. It includes the stages of readiness for change, such as realizing the need for stress reduction (awareness), learning the benefits of stress reduction for reproduction (evaluation) and searching for methods to start with stress (planning). The scale consists of 3 sub-dimensions, namely "Hope and Awareness", "Positive Emotions and Thoughts", "Ready Body and Brain", and a total of 23 items. Since the scale has a positive sentence structure, it allows women to measure their readiness without having negative experiences related to fertility problems in their consciousness and subconscious.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Duzce University, Merkez, Düzce
  - Duzce University, Düzce, Konuralp

IPD SHARING:
Plan to Share IPD: No